CLINICAL TRIAL: NCT05148377
Title: UFH is the Most Used Anticoagulant in Hemodialysis, Decreasing the Risk of Clot Formation in the Circuit.
Acronym: HEPIRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EF101
Record Dates: First submitted 2019-12-26; First posted 2021-12-08 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2020-01

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Parallel clinical study, randomized, double-blind, systematic sampling that evaluated the safety of the sadistic Heparin tested.
Who Masked: Participant, Investigator
Masking Description: The pharmaceutical presentation of the medication to be studied is: solution for injection packaged in 5ml vial and 0.25ml ampoule. All doses have been prepared prior to administration to patients by the LAL Clinic Pharmacy which knows the randomization of the study. It is preparation consisted of preparing the dose of each patient previously calculated based on the weight of each patient and the pharmaceutical presentation of the product randomized into standard 3 ml syringes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium heparin (Heptar) (Experimental): Sodium heparin (Heptar®) produced by Eurofarma Laboratory,
  Interventions: Drug: Heptar
- Liquemine® (Active Comparator): Roche Lab's Liquemine®
  Interventions: Drug: Liquaemin

INTERVENTIONS:
Drug: Liquaemin — The standardized dose for the study was 150UI / kg heparin. It was administered directly through the dialysis equipment.
  Arms: Liquemine®
Drug: Heptar — The standardized dose for the study was 150UI / kg heparin. It was administered directly through the dialysis equipment.
  Other Names: Sodium heparin
  Arms: Sodium heparin (Heptar)

SUMMARY:
The objective of this study was to verify the clinical non-inferiority of the pharmacodynamic effects and the safety of use of the drug Heptar® manufactured by Eurofarma Laboratory, compared to the drug Liquemine®, manufactured by by Roche Laboratory in patients with renal failure undergoing hemodialysis treatment

DETAILED DESCRIPTION:
Parallel clinical study, randomized, double-blind, systematic sampling that evaluated the safety of the sadistic Heparino tested. The study was conducted with the participation of 110 chronic renal failure patients of both sexes. over 18 years old who are undergoing hemodialysis treatment 3 times a week and who fit inclusion and exclusion criteria. The investigational products properly patients were administered during 12 consecutive treatment sessions. Hemodialysis at a dose of 150 IU per kg of weight. The study patients were followed clinically and on a laboratory basis in all hemodialysis sessions according to criteria established by the protocol for verifying the safety in use of the product in study.

The evaluation parameters are:

* Pharmacodynamic effect curve (activity) of heparin verified by dosing of TYPE and anti-Xa markers.
* Effectiveness in maintaining blood coagulation during hemodialysis.

  * Blood loss by coagulation of the system;
  * Blood clotting and venous capillary loss;
  * Trunk of the capillary diolysor in the 12 follow-up sessions.
* Safety in drug use through event monitoring complicating the use of heparin as:

  * Increased hematocrit of the patient;
  * Thrombocytopenia;
  * Bruise;
  * Fever;
  * Reactions to allergic agents;

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of color or social class;
* Age over 18 years, with good clinical characteristics at medical discretion;
* Research patients who agree to participate in the study and sign the consent form free and informed;
* Chronic renal failure patients on dialysis regimen (3 times a week).
* Chronic Kidney Failure with indication for anticoagulant during dialysis

Exclusion Criteria:

* Not agreeing with the terms described in the informed consent;
* Research patients with sensitivity to sadistic heparin;
* Research patients with hypersensitivity to benzyl alcohol;
* Research patients with a history of bleeding or disease that change in coagulation may worsen or terminate the clinical picture, such as ulcer gastric;
* Research patients with a history of peptic ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Blood loss due to system coagulation during 4 weeks of hemodialysis | 4 weeks
  Evaluation of the change of the useful volume of the system below
Loss of venous capillary by clot formation during 4 weeks of hemodialysis | 4 weeks
  Absolut difference of dialyzer lost between the two groups of treatment in the 12 hemodialysis sessions
Change of the useful volume of the system in the dialyzer (priming of dialyzer) | 4 weeks
  Occurrence of events related to the reduction of the useful volume of the system below 80% by thrombus formation in the dialyzer in the 12 hemodialysis sessions

IPD SHARING:
Plan to Share IPD: No